CLINICAL TRIAL: NCT02801604
Title: Attentin® in Children and Adolescents With ADHD - A Non-interventional Study
Acronym: Attention
Status: Completed | Type: Observational
Sponsor: Medice Arzneimittel Pütter GmbH & Co KG (Industry)
Collaborators: University Hospital, Essen (Other)
Responsible Party: Sponsor
Other Study IDs: Attention
Record Dates: First submitted 2016-06-02; First posted 2016-06-16 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2019-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The practicality of most ADHD medications is not or only moderately examined under long term routine conditions. Therefore, in this multi-centre, multi-national prospective non-interventional study, a recommended follow-up time of 12 months will investigate the course of the therapy in children and adolescents with ADHD with prior MPH treatment and their medication change to dexamfetamine in several European countries under daily routine.

It consists of a baseline visit under MPH or another ADHD drug therapy, a change to dexamfetamine, the prospective description of the titration phase and a 12 month maintenance phase. Data on the use of dexamfetamine in routine clinical practice will be collected to describe how dexamfetamine is prescribed, titrated and used in the population of ADHD patients and how these factors influence the general intensity of ADHD and safety events. This study will collect real world data of dexamfetamine and compare descriptively the general intensity of ADHD according to ADHD classification and the impairment due to ADHD under therapy with dexamfetamine to the general intensity of ADHD according to ADHD classification and the impairment due to ADHD under the prior therapy with MPH. Furthermore the utilization of dexamfetamine will be assessed with regards to treatment persistence, compliance, proportion of patients discontinuing treatment and reason for discontinuation. Due to the fact that patients will be treated according to local medical practice it is possible that medication will be changed during the observation period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 6 to 17.11 years
* Current MPH therapy insufficient
* ADHD was classified according to a validated classification system (e.g. DSM or ICD-10)
* No contraindication against dexamfetamine

Exclusion Criteria:

* Contraindication against dexamfetamine

Ages: 6 Years to 215 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents (Age ≥ 6 to 17.11 years) with ADHD, who were treated with methylphenidate (MPH) in the past and, when response to previous MPH treatment is considered clinically inadequate, will be treated with dexamfetamine in this non-interventional study. ADHD was classified according to a classification system of the DSM or ICD and the patient should have no contraindication against dexamfetamine.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-06; Primary Completion 2019-11 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
ADHD classification | baseline until 1st follow-up visit after 6 months
  change from baseline under MPH therapy to the 1st follow-up visit after 6 months under dexamfetamine, assessment by ADHD Rating Scale IV

SECONDARY OUTCOMES:
ADHD classification subgroup: Age | baseline until 1st follow-up visit after 6 months
  change from baseline to 1st follow-up in subgroup of age in years
ADHD classification subgroup: Dose under MPH therapy | baseline until 1st follow-up visit after 6 months
  change from baseline to 1st follow-up in subgroup of MPH dose in mg
ADHD classification subgroup: Dose under dexamfetamine therapy | baseline until 1st follow-up visit after 6 months
  change from baseline to 1st follow-up in subgroup of dexamfetamine dose in mg
ADHD classification subgroup: Baseline ADHD classification | baseline until 1st follow-up visit after 6 months
  change from baseline to 1st follow-up in subgroup baseline ADHD classification, assessment by ADHD Rating Scale IV
Dose-response relationship between dose under dexamfetamine and ADHD classification at 1st follow-up | at 1st follow-up visit, 6 months after baseline
ADHD classification change from baseline to titration and from baseline to 2nd follow-up after 1 year under dexamfetamine | baseline until 2nd follow-up visit after 1 year of examination
  Assessment by ADHD Rating Scale IV
Subscales hyperactivity/impulsivity | baseline until 2nd follow-up visit after 1 year of examination
  Assessment by ADHD Rating Scale IV
Subscales inattention | baseline until 2nd follow-up visit after 1 year of examination
  Assessment by ADHD Rating Scale IV
Response rate, relative reduction in ADHD classification from baseline to 1st follow-up of 30% or more | baseline until1st follow-up visit after 6 months
Overall impairment of the patient's everyday life and disability due to ADHD concerning home life | baseline until 2nd follow-up visit after 1 year of examination
  Assessment for home life
Overall impairment of the patient's everyday life and disability due to ADHD concerning friendships | baseline until 2nd follow-up visit after 1 year of examination
  Assessment for friendships
Overall impairment of the patient's everyday life and disability due to ADHD concerning classroom learning | baseline until 2nd follow-up visit after 1 year of examination
  Assessment for classroom learning
Overall impairment of the patient's everyday life and disability due to ADHD concerning leisure activities | baseline until 2nd follow-up visit after 1 year of examination
  Assessment for leisure activities
Compliance of last MPH intake | baseline
  estimated in per cent
Compliance of last ADHD medication intake (other than MPH) | baseline
  estimated in per cent
Compliance of dexamfetamine intake | titration until 2nd follow-up visit after 1 year of examination
  estimated in per cent
Adverse Drug Reactions under ADHD medication, assessment of blood pressure in mmHg | baseline until 2nd follow-up visit after 1 year of examination
  Assessment of vital parameter: blood pressure in mmHg
Adverse Drug Reactions under ADHD medication, assessment of pulse in beats/min | baseline until 2nd follow-up visit after 1 year of examination
  Assessment of vital parameter: pulse in beats/min
Adverse Drug Reactions under ADHD medication, assessment of weight in kg | baseline until 2nd follow-up visit after 1 year of examination
  Assessment of vital parameter: weight in kg
Adverse Drug Reactions under ADHD medication, assessment of height in cm | baseline until 2nd follow-up visit after 1 year of examination
  Assessment of vital parameter: height in cm

CONTACTS AND LOCATIONS:
Overall Officials: Michael Huss, Prof. Dr., Principal Investigator — Child and Adolescent Psychiatry, University of Medicine, Mainz, Germany
Locations (1):
- Child and Adolescent Psychiatry, University of Medicine, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No